CLINICAL TRIAL: NCT04232618
Title: Field Evaluation of a Point-of-care Triage Test for Active Tuberculosis
Brief Title: Point-of-care Triage Test for Active Tuberculosis
Acronym: TriageTB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Makerere University (Other); Find (Other); Leiden University Medical Center (Other); Medical Research Council Unit, The Gambia (Other); LINQ Management GMBH (Unknown)
Responsible Party: Principal Investigator, Prof Gerhard Walzl, Executive Head of Department of Biomedical Sciences, University of Stellenbosch
Other Study IDs: RIA2018D-2499
Record Dates: First submitted 2019-11-26; First posted 2020-01-18 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Finger stick capillary blood for POC test strip, Serum collection and storage, Whole blood collection for isolation of peripheral blood mononuclear cells (PBMCs), PAXgene collection for storage of mRNA, Sputum for testing and storage, Urine for storage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FIND cohort: Evaluation of biomarkers in serum samples from 500 people with suspected TB from non-African countries provided by FIND diagnostic biorepository.
- Phase 1: Evaluate the basic 3-marker multi-biomarker test (MBT) signature in 150 participants across three African sites. This will be used to lock down the final MBT signature to be used in the next phase of testing.
  Interventions: Diagnostic Test: Multi-biomarker point-of-care test
- Phase 2: Enrolment of 750 participants across three African sites using the locked down MBT signature from phase 1.
  Interventions: Diagnostic Test: Multi-biomarker point-of-care test

INTERVENTIONS:
Diagnostic Test: Multi-biomarker point-of-care test — Lateral flow device containing a combination of markers which have been shown to be associated with active tuberculosis.
  Groups: Phase 1; Phase 2

SUMMARY:
Background:

Tuberculosis (TB) is a bacterial lung infection leaving 3.6 million people undiagnosed each year. Thirty percent of infected people do not receive treatment due to failure to receive diagnostic testing or being lost to follow-up between testing and availability of results.

Objective:

To refine and field-validate a point-of-care (POC) finger stick blood test for use worldwide to triage for active TB.

Eligibility:

Persons aged 12 - 70 years with symptoms suggestive of TB disease

Study design:

Participants will be screened with:

Medical history Physical exam HIV test, diabetes screening Blood (finger stick and venous), sputum and urine collection Chest X-ray TB positive participants will receive treatment from the National TB Program at Community Health Centres and clinics.

DETAILED DESCRIPTION:
This study aims to make widely available an inexpensive, easy to use point-of-care finger stick test to triage patients presenting with signs and symptoms consistent with active TB. From previous experience in EDCTP-funded studies, approximately 30% of such patients test positive for TB, with the vast majority having respiratory illnesses other than active TB, including acute upper or lower respiratory tract infections or exacerbations of chronic obstructive pulmonary disease. The proposed finger stick test is designed, with the aim of use, as a TB rule out test such that resources required for further testing can be used with more efficiency.

The majority (60%) of suspected TB cases are seen at public health facilities, however many facilities in high TB prevalence areas still do not have access to efficient TB diagnostic services due to logistical and financial constraints that plague these settings. Currently available diagnostics include radiological and microbiological testing, though each has drawbacks for use in primary care facilities.

The TriageTB consortium will be evaluating combinations of biomarkers in samples from African and Non-African individuals suspected of having TB in order to identify the optimal biomarker signature for global identification of patients with high likelihood of TB. A device has been developed, which measures a combination of biomarkers in finger stick capillary blood and has been validated in the laboratory setting. Previous EDCTP-funded projects identified a promising 6-marker biosignature which has been shown to have potential for being reduced to a 3- or 4- marker signature. The 3-marker signature has the added benefit of potential for treatment monitoring applications. A triage test as proposed here would significantly speed up and streamline diagnostic approaches in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 to 70 years.
2. Symptoms suggestive of TB disease: cough for ≥ two weeks plus at least one of the following: fever, malaise, weight loss, night sweats, haemoptysis, chest pain or loss of appetite.
3. Participants aged ≥18 years-old: Willing to give informed consent to take part in the study, including

   1. Willingness to undergo HIV testing and be willing to have their HIV infection status disclosed to the study field workers.
   2. Willingness to have study samples stored indefinitely.
4. Participants aged ≥12 and <18 years:

   1. Accompanied by a parent or legal guardian/caregiver/representative who is willing to provide informed consent for study procedures as above, and
   2. The child is willing to give informed assent for study procedures as above and the attending research staff member is satisfied that the participant understands the study satisfactorily.

Participants who had previous TB, extra-pulmonary TB in addition to pulmonary TB, drug resistance detected on GeneXpert® Ultra or culture, or other concomitant diseases will not be excluded from enrolment. People living with, and without, HIV will be enrolled.

Exclusion Criteria:

1. Stable permanent residence in study area for less than 3 months; no permanent address or planned relocation in the next six months.
2. Pregnancy or breastfeeding.
3. Hb < 9g/l.
4. Current systemic steroid use or immune suppression therapy in the past four weeks.
5. On TB treatment or Isoniazid Preventive Treatment (IPT) currently or in the last ninety days.
6. Known quinolone or aminoglycoside antibiotic use reported in the past 60 days.
7. Participants aged ≥18 years-old: Unable to provide informed consent (eg due to mental impairment), or are deemed by the attending research staff member as unable to complete study procedures (eg. due to substance abuse affecting the participant's level of function).
8. Participants aged ≥12 and <18 years:

   1. Either the parent/guardian is willing to give informed consent or the participant is unwilling to give informed assent.
   2. Both the parent/guardian and the child are willing to provide consent and assent, but in the attending researcher's opinion there is a problem with the validity of the consent (eg. because of suspected mental impairment) or with completion of study procedures (eg. because of substance abuse of parent or child).

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are recruited from known TB endemic areas across three African countries.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Global diagnostic bio-signature for diagnosing active TB | 4 years
  Accuracy of a point-of-care multi-biomarker test (POC-MBT) in active, pulmonary tuberculosis.

SECONDARY OUTCOMES:
Use of MBT for treatment response | 4 years
  Accuracy of the point-of-care multi-biomarker test as an indicator of tuberculosis treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Walzl, MBCHB; PhD, Principal Investigator — University of Stellenbosch
Locations (1):
- Stellenbosch University, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suliman S, Thompson EG, Sutherland J, Weiner J 3rd, Ota MOC, Shankar S, Penn-Nicholson A, Thiel B, Erasmus M, Maertzdorf J, Duffy FJ, Hill PC, Hughes EJ, Stanley K, Downing K, Fisher ML, Valvo J, Parida SK, van der Spuy G, Tromp G, Adetifa IMO, Donkor S, Howe R, Mayanja-Kizza H, Boom WH, Dockrell HM, Ottenhoff THM, Hatherill M, Aderem A, Hanekom WA, Scriba TJ, Kaufmann SHE, Zak DE, Walzl G; GC6-74 cohort study team, The ACS cohort study team. Four-Gene Pan-African Blood Signature Predicts Progression to Tuberculosis. Am J Respir Crit Care Med. 2018 May 1;197(9):1198-1208. doi: 10.1164/rccm.201711-2340OC. PMID 29624071
- [Background] Tadesse T, Demissie M, Berhane Y, Kebede Y, Abebe M. Two-thirds of smear-positive tuberculosis cases in the community were undiagnosed in Northwest Ethiopia: population based cross-sectional study. PLoS One. 2011;6(12):e28258. doi: 10.1371/journal.pone.0028258. Epub 2011 Dec 2. PMID 22164256
- [Derived] Richardson TR, Smith B, Malherbe ST, Shaw JA, Noor F, MacDonald C, van der Spuy GD, Stanley K, Carstens A, Fisher TL, van Rensburg I, Flinn M, Snyders C, Johnson I, Fransman B, Dockrell H, Thwaites G, Thuong NTT, Schacht C, Mayanja-Kizza H, Nsereko M, Tjon Kon Fat EM, Corstjens PLAM, Geluk A, Ruhwald M, Penn-Nicholson A, Chegou NN, Sutherland J, Walzl G; TrENDx consortium. Field evaluation of a point-of-care triage test for active tuberculosis (TriageTB). BMC Infect Dis. 2023 Jul 3;23(1):447. doi: 10.1186/s12879-023-08342-5. PMID 37400753
- See also: TB Statistics for South Africa — http://tbfacts.org/tb-statistics-south-africa/